CLINICAL TRIAL: NCT01219907
Title: Phase I Study of Adoptive T-Cell Therapy With HER-2/Neu (HER-2)-Specific Memory CD8+ T Lymphocytes Obtained Following In Vivo Priming With a Peptide Vaccine in Patients With Advanced Stage HER-2-Positive Breast Cancer
Brief Title: Ex Vivo-Expanded HER2-Specific T Cells and Cyclophosphamide After Vaccine Therapy in Treating Patients With HER2-Positive Stage IV Breast Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Salazar, Lupe, Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7266; NCI-2010-01792
Record Dates: First submitted 2010-09-22; First posted 2010-10-13 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: HER2-positive Breast Cancer; Male Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — Cyclophosphamide; Flow Cytometry; Immunoenzyme Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm I (Experimental): VACCINE THERAPY: Patients receive HER2 peptide vaccine intradermally once weekly for 3 weeks.
  CHEMOTHERAPY: Patients receive cyclophosphamide IV on day -1.
  IMMUNOTHERAPY: Patients receive ex vivo-expanded HER2 specific T-cell IV over 30 minutes on days 1, 10, and 20.
  Interventions: Biological: HER-2/neu peptide vaccine; Drug: cyclophosphamide; Biological: ex vivo-expanded HER2-specific T cells; Other: laboratory biomarker analysis; Other: flow cytometry; Other: immunoenzyme technique

INTERVENTIONS:
Biological: HER-2/neu peptide vaccine — Given intradermally
  Other Names: HER-2
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana; Enduxan
Biological: ex vivo-expanded HER2-specific T cells — Given IV
Other: laboratory biomarker analysis — Correlative studies
Other: flow cytometry — Correlative studies
Other: immunoenzyme technique — Correlative studies
  Other Names: immunoenzyme techniques

SUMMARY:
RATIONALE : Laboratory-treated T cells may stimulate the immune system in different ways and stop tumor cells from growing. Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Vaccines made from HER2 peptides may help the body build an effective immune response to kill tumor cells that express HER2. Giving laboratory-treated T cells and cyclophosphamide after vaccine therapy may be an effective treatment for breast cancer.

PURPOSE: This phase I trial is studying the side effects and best dose of ex vivo-expanded HER2-specific T cells when given together with cyclophosphamide after vaccine therapy in treating patients with HER2-positive stage IV breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the feasibility of expanding HER-2-specific effector T cells (TE) ex vivo from CD62L+ TCM and CD62L- TEM from patients immunized with a HER-2 peptide vaccine.

II. To evaluate the safety of infusing autologous ex vivo expanded HER-2-specific T cells into patients with advanced HER-2+ breast cancer.

SECONDARY OBJECTIVES:

I. To evaluate the persistence, function, and phenotype of adoptively transferred HER-2-specific TE cells derived from TCM or TEM precursors.

II. To investigate the potential anti-tumor effects of therapy with ex vivo expanded HER-2-specific T cells in patients with advanced HER-2+ breast cancer.

OUTLINE : This is a dose-escalation study of ex vivo-expanded HER2-specific T cells.

VACCINE THERAPY: Patients receive HER2 peptide vaccine intradermally once weekly for 3 weeks.

CHEMOTHERAPY: Patients receive cyclophosphamide IV on day -1.

IMMUNOTHERAPY: Patients receive ex vivo-expanded HER2 specific T-cell IV over 30 minutes on days 1, 10, and 20.

After completion of study treatment, patients are followed up on days 28, 35, 49, 63 and then monthly thereafter for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HER-2+ Stage IV breast cancer that have been maximally treated and not in a complete remission
* Subjects must be > 18 years old
* Extra skeletal disease that can be accurately measured in at least one dimension as >= 20 mm with conventional CT techniques or >= 10 mm with spiral CT scan
* Skeletal or bone-only disease that is measurable by FDG PET imaging will also be allowed
* Patients can be receiving trastuzumab and/or hormonal therapy and/or bisphosphonates
* HER2 overexpression in the primary tumor or metastasis by IHC of 2+ or 3+, or documented gene amplification by FISH analysis; if over expression is 2+ by IHC, patients must have HER2 gene amplification documented by FISH
* Performance Status Score (ECOG/Zubrod Scale) must be =< 2
* Patients must be off all immunosuppressive treatments such as chemotherapy or systemic steroid therapy a minimum of 3 weeks prior to initiation of study (i.e. first vaccination)
* Patients on trastuzumab must have a baseline LVEF measured by MUGA or echocardiogram >= the lower limit of normal for the facility within 3 months of enrollment to study
* Subjects must be HLA-A2 (HLA A*0201) positive
* ANC >= 1000/mm^3
* Hgb >= 10 mg/dl
* Platelet count >= 75,000/mm^3
* Men and women of reproductive ability must agree to use contraceptives during the entire study period

Exclusion Criteria:

* Serum creatinine > 2.0 mg/dl
* Serum bilirubin > 2.5 times the upper limit of normal
* Contraindication to receiving GM-CSF based vaccine products
* New York Heart Association functional class III-IV heart failure, symptomatic pericardial effusion, or unstable angina
* History of disorders associated with immunosuppression such as HIV
* Pregnant or breast-feeding women
* ANC < 1000/mm^3
* Hgb < 10 mg/dl
* Platelet count < 75,000/mm^3
* Active brain metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Ability to expand HER-2-specific T cells ex vivo from memory T cell subsets which are derived from patients with advanced HER-2 expressing cancer | After leukapheresis (2 weeks after 3rd vaccination) and prior to chemotherapy
  Ability to expand HER-2-specific T cells ex vivo from memory T cell subsets which are derived from patients with advanced HER-2 expressing cancer will be defined as feasible if the minimum target expansion of HER-2-specific T cells is achieved in ≥2/3 expansions in ≥7/10 subjects.
Safety and systemic toxicity as assessed at regular time points by NCI common toxicity criteria (CTCAE v 4.0). Stopping rules for the study protect patients against therapy with a rate of severe toxicity of 20% or greater. | At week 1, 2, 3, post T-Cell infusion day 1, 10, 20, 28, 35, 49, 63, then every 3 months for a year.

SECONDARY OUTCOMES:
Extent to which to HER-2-specific T cell immunity can be boosted successfully with adoptive immunotherapy will be defined by quantitative assessment of HER-2-specific CD8+ T cells assessed by cytokine flow cytometry (CFC), Elispot, and tetramer staining | Post T-Cell-infusion on day 10, 20, 28, 35, 49, 63, then monthly for one year.
Persistence of T cell immune augmentation in vivo after adoptive transfer of HER-2-specific T cells as assessed by presence of HER-2-specific central memory T cells and effector memory T cells | Every month for 1 year following the last infusion
Anti-tumor effects of HER-2-specific T cells as assessed by RECIST criteria | Day 63 post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Lupe Salazar, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States